CLINICAL TRIAL: NCT01772914
Title: Copeptin During a Standardized Oral Glucose Tolerance Test and a Mixed Meal Tolerance Test
Brief Title: Copeptin Changes After Food Intake
Acronym: CoMeal
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Mirjam Christ-Crain, Prof. Dr. med., University Hospital, Basel, Switzerland
Other Study IDs: CoMeal 2013
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Adults; Copeptin
Keywords: Copeptin; eating; glucose tolerance test; mixed meal test; physiological
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Serum EDTA
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether copeptin levels are affected by food intake.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years

Exclusion Criteria:

* Intake of any kind of medication (except birth control pill)
* BMI >30 kg/m2
* Evidence of any acute illness
* History of chronic illness
* Pregnancy
* Known galactosemia or maltose malabsorption
* Baseline glucose level >5.5 mmol/l Baseline sodium level <135 mmol/l or >145 mmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes in copeptin levels after intake of a oral glucose tolerance test- and a mixed meal tolerance test liquid | 30, 60, 90, 120, 180 minutes after intake of the test liquids

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof.Dr.med., Principal Investigator
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Walti C, Siegenthaler J, Christ-Crain M. Copeptin levels are independent of ingested nutrient type after standardised meal administration--the CoMEAL study. Biomarkers. 2014 Nov;19(7):557-62. doi: 10.3109/1354750X.2014.940504. Epub 2014 Sep 16. PMID 25224842